CLINICAL TRIAL: NCT00716794
Title: A Phase I/II, Open-Label, Dose Ranging Study of the Safety, Tolerance, Pharmacokinetics and Potential Activity of HE3235 When Administered Orally to Patients With Prostate Cancer
Brief Title: A Phase I/II Study of HE3235 in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Harbor Therapeutics (Industry)
Responsible Party: Nanette Onizuka-Handa/Sr. Vice President, Regulatory Affairs and Quality, Harbor BioSciences, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE3235-0201
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; HE3235; Apoptone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 17-ethynylandrostane-3,17-diol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: HE3235 — HE3235 will be administered orally in 28 day cycles.
  Other Names: Apoptone

SUMMARY:
This is a phase I/II, open-label, dose escalation study of HE3235 administered orally to patients with advanced prostate cancer who have failed hormone therapy and at least one taxane based chemotherapy regimen.

ELIGIBILITY:
Main Inclusion Criteria:

* Patient is male and at least 18 years of age, at the time of screening;
* Patient has metastatic disease (any T, any N, M1);
* Patient has failed at least 1 taxane regimen; or Patient has symptomatic or asymptomatic CRPC and is chemotherapy-naïve
* Patient has histologically or cytologically confirmed adenocarcinoma of the prostate;
* Patient has progression of disease despite adequate hormone therapy, demonstrated by one of the following:

  * PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions, at least 1 week apart.
  * Evaluable disease progression by modified RECIST (Response Evaluation Criteria in Solid Tumors) criteria;
  * Progression of metastatic bone disease on bone scan with > 2 new lesions
* Patient has ECOG (Eastern Cooperative Oncology Group) performance status of 0-2;

Main Exclusion Criteria:

* Patient has symptomatic parenchymal brain metastases or active epidural disease requiring whole-brain irradiation Treated epidural disease is allowed
* Patient has active infection;
* Patient having a history of clinically significant cardiovascular disease (such as CHF), clinically significant hepatic, respiratory or renal abnormalities;
* Patient who has any clinically significant abnormalities in laboratory results at screening
* Patient who has a history of clinically significant neurological or psychiatric condition;

Additional criteria are applicable to expansion cohorts.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerance of HE3235 when administered orally to prostate cancer patients in 28 day cycles. | Treatment period
To evaluate the pharmacokinetic profiles of HE3235 and major metabolites at different dose levels after 28 days of dosing. | Treatment period
To assess potential activity of HE3235 in prostate cancer patients. | Treatment period and post-study follow-up period

SECONDARY OUTCOMES:
Explore circulating tumor cell (CTC) enumeration in response to treatment as a marker evaluating whether an investigational therapy is effective for tumor treatment | Treatment period
Evaluate the role of molecular profiling of CTC in predicting sensitivity to treatment and treatment response. | Treament period and post-study follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Stickney, MD, Study Director — Harbor Therapeutics
Locations (8):
- United States (8):
  - Scottsdale, Arizona
  - Encinitas, California
  - Roseville, California
  - San Francisco, California
  - New York, New York
  - Charlotte, North Carolina
  - San Antonio, Texas
  - Seattle, Washington